CLINICAL TRIAL: NCT05000294
Title: Atezolizumab Plus Tivozanib in Immunologically Cold Tumor Types
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: interim analysis
Sponsor: University of Florida (Other)
Collaborators: Genentech, Inc. (Industry); Aveo Oncology Pharmaceuticals (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UF-STO-ETG-003; OCR40357 (Other: University of Florida); IRB202101773 (Other: University of Florida IRB-01)
Record Dates: First submitted 2021-08-10; First posted 2021-08-11 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Bile Duct Cancer; Gall Bladder Cancer; Breast Cancer; Neuroendocrine Tumors; Ovarian Cancer; Pancreatic Adenocarcinoma; Soft Tissue Sarcoma; Vulvar Cancer; Prostate Cancer
Keywords: immunologically cold tumors; breast cancer; bile duct cancer; gallbladder cancer; neuroendocrine cancer; ovarian cancer; pancreatic adenocarcinoma; soft tissue sarcoma; prostate cancer; vulvar cancer; TKI; checkpoint inhibitor
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms; Breast Neoplasms; Neuroendocrine Tumors; Ovarian Neoplasms; Sarcoma; Vulvar Neoplasms; Prostatic Neoplasms; Carcinoma, Neuroendocrine | interventions — atezolizumab; tivozanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Atezolizumab + Tivozanib (Experimental)
  Interventions: Drug: Atezolizumab; Drug: Tivozanib

INTERVENTIONS:
Drug: Atezolizumab — Subjects on both the phase Ib and phase II portions of this study will receive 1680 mg intravenously of atezolizumab on Day 1 of each 28 day cycle.
  Other Names: Tecentriq
Drug: Tivozanib — Subjects in both the phase Ib and phase II portions of the study will take tivozanib orally once daily on Days 1-21 of each 28 day cycle. Subjects on the phase Ib will be assigned to receive either 1.34 mg/day (Dose level 0) or 0.89 mg/day (Dose level -1). Subjects in the phase II portion of the study will receive 0.89 mg/day.
  Other Names: Fotivda

SUMMARY:
Checkpoint inhibitor therapy represents a significant advance in cancer care. The interaction between PD-1 and PD-L1 induces immune tolerance, and the inhibition of this interaction is an effective treatment strategy for numerous malignancies.

Despite its demonstrated potential, immunotherapy is not currently thought to be an effective intervention in the treatment of several immunologically "cold" tumors such as prostate cancer, biliary tract cancers, soft tissue sarcomas, well-differentiated neuroendocrine tumors, microsatellite stable colorectal cancer, pancreatic cancer, and non-triple negative breast cancer.

Vascular endothelial growth factor (VEGF) is thought to play a key role in modulating the anti-tumor immune response. Vascular endothelial growth factor (VEGF) is secreted by tumors and leads to endothelial cell proliferation, vascular permeability, and vasodilation. This in turn leads to the development of an abnormal vasculature with excessive permeability and poor blood flow, limiting immune surveillance. In addition, VEGF inhibits dendritic cell differentiation, limiting the presentation of tumor antigens to CD4 and CD8 T cells. Vascular endothelial growth factor (VEGF). VEGF tyrosine kinase inhibitors (TKIs) VEGF-TKIs are currently utilized in the treatment of a variety of malignancies and are widely utilized in combination with checkpoint blockade in the treatment of clear cell kidney cancer.

Through the inhibition of VEGF, it may be possible to potentiate the effect of immune checkpoint blockade even in tumors which have traditionally been thought to be unresponsive to immunotherapy. This study aims to evaluate the combination of the immune checkpoint inhibitor atezolizumab and the VEGF-TKI tivozanib in a variety of tumors which have a low response rate to checkpoint inhibitor therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have had at least one prior treatment with systemic therapy for advanced and unresectable, or metastatic disease OR is intolerant to, has refused or for whom there are no standard therapies that impart significant clinical benefit in the opinion of the treating investigator.
* An Eastern Cooperative Oncology Group (ECOG) Performance Status less than or equal to 1 for phase 1B. An ECOG Performance Status less than or equal to 2 for phase 2.
* Subjects must not have more than one malignancy at the time of enrollment
* Adult subjects ≥ eighteen years of age
* A clinical diagnosis consistent with stage IV "immunogenically cold" or otherwise incurable cancer of one of the following histologies: i) bile duct or gallbladder cancer ii) Metastatic breast cancer, HR-negative HER2-positive, who have received at least 3 lines of therapy for disease progression that includes: trastuzumab, pertuzumab/trastuzumab, and ado-trastuzumab emtansine iii) neuroendocrine cancer with the following pathological characteristics: grade 2 or 3; well- or moderately- differentiated (Grades 1, 4, and poorly differentiated neuroendocrine pathologies are not eligible) iv) FIGO stage IV or metastatic (using 2021 FIGO classification) high grade serious or high grade endometrioid (based on local histopathological findings) ovarian cancer, primary peritoneal cancer and / or fallopian-tube cancer that is platinum resistant, with no acceptable standard of care v) pancreatic adenocarcinoma vi) soft tissue sarcoma vii) prostate cancer subjects who are castrate-resistant (testosterone ≤ 50 ng/dL) and have progressed on, declined, or are intolerant to other standard of care therapies. Subjects with prostate cancer must have failed at least one line of treatment with an androgen inhibitor (AI) (i.e. enzalutamide, abiraterone, etc.) or cytotoxic chemotherapy in the advanced or metastatic setting viii) vulvar cancer
* Adequate hematologic and end-organ function
* Subjects receiving therapeutic anticoagulation must be on a stable anticoagulant regimen for ≥ 2 weeks at start of protocol treatment
* Negative hepatitis B surface antigen (HBsAg) test at screening
* Negative HIV test at screening with the following exceptions: subjects with a positive HIV test at screening are eligible only if they meet the following three conditions: 1) Are stable on anti-retroviral therapy 2) Have a CD4 count ≥ 200/uL AND 3) Have an undetectable viral load.
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception (with a failure rate of <1% per year) to avoid pregnancy throughout the study and for at least 160 days after the last dose of either study drug to minimize the risk of pregnancy.
* Males with female partners of child-bearing potential must agree to use physician-approved contraceptive methods throughout the study and should avoid conceiving children for 160 days following the last dose of study drug.
* Measurable disease by RECIST criteria
* A life expectancy of ≥ 12 weeks
* Written informed consent obtained from the subject and the subject agrees to comply with all the study-related procedures
* Must have formalin-fixed paraffin embedded (FFPE) tissue or 12 unstained slides available for research purposes. Tissue must have been obtained within the last 3 years.
* If a new biopsy is needed for diagnostic reasons, the biopsy must be performed from a tumor site that is not the only site of measurable disease
* Subject must be able to swallow capsules

Exclusion Criteria:

* Subjects with known MSI-H or dMMR tumor status
* Subjects with severe uncontrolled hypertension as defined as systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg
* Subjects who have had prior treatment with vascular endothelial growth factor receptor (VEGFR) tyrosine kinase inhibitors
* Females or males of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 160 days after the last dose of study drug
* Females who are pregnant or breastfeeding
* History of leptomeningeal disease
* Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN)
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently, except in the case of ovarian cancer with ascites, which may require more frequent drainage). Subjects with indwelling catheters are allowed.
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

  1. subjects with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
  2. subjects with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
  3. subjects with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., subjects with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

     * Rash must cover <10% of body surface area
     * Disease is well controlled at baseline and requires only lowpotency topical corticosteroids
     * There has been no occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Active tuberculosis
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* History of malignancy other than the malignancies listed in the inclusion criteria of enrollment within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer
* Severe infection within 4 weeks prior to initiation of study treatment including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia, or any active infection that could impact patient safety
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment. Note: Subjects receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
* Prior allogeneic stem cell or solid organ transplantation
* Current treatment with anti-viral therapy for hepatitis B virus (HBV)
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
* Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

  1. Subjects who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study.
  2. Subjects who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* History of any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician
* Administration of a vaccine containing live virus within 30 days prior to the first dose of trial treatment, during treatment with atezolizumab, and for 160 days after the last dose of atezolizumab. Note: Most flu vaccines are killed viruses, with the exception of the intra-nasal vainer (Flu-Mist) which is an attenuated live virus and therefore prohibited for 30 days prior to first dose. Subjects may receive non-live COVID-19 vaccine.
* Prisoners or subjects who are involuntarily incarcerated, or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.
* Subjects with Tumor Mutation Burden (TMB) ≥10
* Treatment with any cancer directed therapy (i.e. chemotherapy, radiation therapy, Y90, microwave ablation, immunotherapy, etc.) within 28 days of study start
* Subjects with treated brain metastases that have remained stable for at least 90 days without steroids are allowed. Subjects with signs of symptoms or history of brain metastasis must have a CT or MRI of the brain within 30 days prior to the start of protocol therapy.
* Subjects with autoimmune diseases requiring current treatment and subjects with history of severe autoimmune diseases, subjects with hypothyroidism, adrenal insufficiency, or pituitary insufficiency who are stable on therapy are allowed.
* Inability to discontinue use of medications contraindicated by the study treatment
* Proteinuria > 2.5 g/24 hours or 3+ with urine dipstick
* QTc interval > 470 at screening or known cardiovascular disease defined as (a) a clinically significant abnormal ECG at screening, or (b) myocardial infarction within 12 weeks prior to start of protocol therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 30 months
  To determine the best overall response rate (ORR) of atezolizumab plus tivozanib in subjects with immunologically cold tumors

SECONDARY OUTCOMES:
Progression free survival (PFS) | 30 months
  To determine the progression free survival (PFS) of subjects with immunologically cold tumors receiving atezolizumab plus tivozanib
Overall survival (OS) | 30 months
  To determine the overall survival (OS) of subjects with immunologically cold tumors receiving atezolizumab plus tivozanib.
Disease control rate (DCR) | 30 months
  To determine the disease control rate (DCR) of subjects with immunologically cold tumors receiving atezolizumab plus tivozanib. DCR is defined as percentage of subjects who achieve complete response, partial response and stable disease during the course of study using RECIST v1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Leighton Elliott, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramnaraign BH, Lee JH, Ali A, Rogers SC, Fabregas JC, Thomas RM, Allegra CJ, Sahin I, DeRemer DL, George TJ, Chatzkel JA. Atezolizumab plus tivozanib for immunologically cold tumor types: the IMMCO-1 trial. Future Oncol. 2022 Nov 18. doi: 10.2217/fon-2022-0392. Online ahead of print. PMID 36399037